CLINICAL TRIAL: NCT06587191
Title: Retrospective Non-interventional Study Assessing Efficacy and Safety of Emapalumab in Children With Primary Hemophagocytic Lymphohistiocytosis (pHLH)
Brief Title: Emapalumab Efficacy in Children With Primary Hemophagocytic Lymphohistiocytosis
Acronym: CGM EMA
Status: Active, not recruiting | Type: Observational
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Other Study IDs: NCHPOI-2024--07
Record Dates: First submitted 2024-08-22; First posted 2024-09-19 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-08

CONDITIONS: Primary Hemophagocytic Lymphohistiocytosis
Keywords: primary hemophagocytic lymphohistiocytosis; children; treatment; emapalumab
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this retrospective study is to assess efficacy and safety of emapalumab prescribed for the treatment in children with refractory from of pHLH.

DETAILED DESCRIPTION:
Primary hemophagocytic lymphohistiocytosis (pHLH) encompasses a group of genetically determined disorders, characterized by severe, often fulminant systemic inflammation, cytopenia and multiple organ involvement. The disease manifests predominantly in the early childhood, has high mortality rate and in most cases requires hematopoietic stem cell transplantation (HSCT) as the only currently available curative option. Yet, HSCT outcomes are dependent on the state of remission of the underlying systemic inflammation and infections complications, as well as organ damage due to the side effects of the chemotherapeutic drugs received prior to it. For years the gold standard of HLH treatment has been the dexamethasone and etoposide-based HLH-2004 protocol, yet it failed to uniformly control the disease. An alternative regiment combining antithymocyte globulin and corticosteroids demonstrated good results but barely improved survival. Also, no universally accepted treatment exists for relapsed or refractory hemophagocytic lymphohistiocytosis. Advances in availability of biologic treatments open up new possibilities of HLH therapy, with several targets proposed in recent years. Interleukin 6 inhibitor tocilizumab, interleukin 1 inhibitor anakinra, Janus-kinase inhibitor (JAKinib) ruxolititnib have been used for HLH treatment, with variable results.

Mounting evidence provides support for the pivotal pathogenic role of interferon-γ (IFNg) in hemophagocytic lymphohistiocytosis. Emapalumab is a fully human IgG1 anti-interferon-γ monoclonal antibody that binds free and receptor-bound interferon-γ and inhibits its biologic activity. The data accumulated from the phase II/III clinical trial and reports of the small groups of patients demonstrate its efficacy in pHLL.

The study will collect and analyze information of the effectiveness and safety of emapalumab treatment that was previously prescribed in a cohort of seven pediatric patients with pHLH.

Criteria for inclusion in the study were:

1. age from 0 to 18 y.
2. the diagnosis of pHLH ( established according to the Histiocytic society criteria).
3. treatment with empalumab for at least 2 weeks
4. signed informed consent for participation in the study Exclusion criteria - not applicable.

ELIGIBILITY:
Inclusion Criteria:

Criteria for inclusion in the study were:

1. age from 0 to 18 y.
2. the diagnosis of pHLH ( established according to the Histiocytic society criteria).
3. treatment with empalumab for at least 2 weeks
4. signed informed consent for participation in the study

Exclusion Criteria:

not applicable. signed informed consent for participation in the study

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The disease manifests predominantly in the early childhood, has high mortality rate.
  Also, no universally accepted treatment exists for relapsed or refractory hemophagocytic lymphohistiocytosis. For years the gold standard of HLH treatment has been the dexamethasone and etoposide-based HLH-2004 protocol, yet it failed to uniformly control the disease.
Sampling Method: Probability Sample
Enrollment: 7 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Dynamics of severity clinical and laboratory activity using scale H-score. | at the day the first dose of study treatment was administered, further at days 14, 28 and at the end of treatment, an average 45 days

SECONDARY OUTCOMES:
Adverse events | at the day the first dose of study treatment was administered, further at days 14, 28 and at the end of treatment, an average 45 days
Infection complications before therapy | at the day the first dose of study treatment was administered, further at days 14, 28 and at the end of treatment, an average 45 days
Infection complications after therapy | at the day the first dose of study treatment was administered, further at days 14, 28 and at the end of treatment, an average 45 days

CONTACTS AND LOCATIONS:
Overall Officials: Anna Scherbina, MD,Phd, Study Director — Chief HSCT department at Federal Research Center for pediatric hematology, oncology and immunology
Locations (1):
- Research Institute of Pediatric Hematology, Oncology and Immunology, Moscow, Russia